CLINICAL TRIAL: NCT03998384
Title: Retrobulbar Injection of Autoserum in the Treatment of Retinitis Pigmentosa: A Prospective, Non-randomized Interventional Study
Brief Title: A New Treatment of Retinitis Pigmentosa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHAIER2019IRB01
Record Dates: First submitted 2019-06-07; First posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: Two eyes of one patient with RP will be divided into two groups. One eye with more serious retinal atrophy will receive retrobulbar injection of autoserum, and the other eye will receive retrobulbar injection of saline solution.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group of autoserum (Active Comparator): One of two eyes of one patient which is assessed to have more serious retinal atrophy will receive the retrobulbar injection of autoserum.
  Interventions: Procedure: retrobulbar injection of autoserum
- group of placebo (Placebo Comparator): The other eye which is assessed to have milder retinal atrophy will receive the retrobulbar injection of saline solution.
  Interventions: Procedure: retrobulbar injection of placebo

INTERVENTIONS:
Procedure: retrobulbar injection of autoserum — Retrobulbar block is usually a type of regional anesthetic nerve block used in intraocular surgery. In this technique, local autoserum is injected into the retrobulbar space for the neurotrophic purpose.
  Arms: group of autoserum
Procedure: retrobulbar injection of placebo — Retrobulbar block is usually a type of regional anesthetic nerve block used in intraocular surgery. In this technique, normal saline (NS) is injected into the retrobulbar space as a comparison
  Arms: group of placebo

SUMMARY:
This study is designed to assess and to evaluate the therapeutic effect of retrobulbar injection of autoserum in the treatment of retinitis pigmentosa.

DETAILED DESCRIPTION:
The retinitis pigmentosa(RP) is an hereditary disease which causes visual deficiency leading to blindness. The methods of treatment include gene therapy, stem cell therapy and visual prothesis, etc. But all these methods own limitations can not be conquered in a short period. It was proved that vascular endothelial growth factor (VEGF) and pigment epithelium derived factor (PEDF) decreased in the aqueous humor of patients of RP. But the traditional exogenous nerve growth factors (NGFs) were immunogenic proteins and may cause inflammation. Autoserum contain a large amount of active factors and will not cause exclusive reaction. In this study we aim to assess and to evaluate the therapeutic effect and the safety of retrobulbar injection of autoserum in the treatment of retinitis pigmentosa.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of retinitis pigmentosa

Exclusion Criteria:

* Suspected glaucoma, suspected optic nerve disease, blindness due to other ocular disease
* Combined with serious systemic disease
* Can not cooperate with the interventions and examinations.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of the visual acuity | one day before injection, one day, one month, three months and six months after surgery
  To measure the visual acuity with logarithmic visual chart.
Change of the contrast sensitivity | one day before injection, one month, three months and six months after surgery
  To access the change of contrast sensitivity in different special frequency.
Change of the electrophysiological detection (flash electroretinogram) | one day before injection, three months and six months after surgery
  To evaluate the retinal function with the use of flash electroretinogram (F-ERG).
Change of the electrophysiological detection (electro-oculogram) | one day before injection, three months and six months after surgery
  To evaluate the retinal function with the use of electro-oculogram (EOG)